CLINICAL TRIAL: NCT06031805
Title: a French Observational Prospective Multicenter Study of Adult Patients Treated in the Real-life Setting With Olaparib for the Treatment of Metastatic Castration-resistant Prostate Cancer
Brief Title: PRostate Olaparib Real World Evidence Study
Acronym: PROWESs
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0817R00049
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This French non-interventional prospective multicenter cohort study is conducted to study the added value of olaparib in the treatment of patients with mCRPC in the real world setting in terms of treatment sequencing, effectiveness, safety and BRCA testing patterns and thus inform future clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult male patients (≥ 18 years old)
* With metastatic castration-resistant prostate cancer - Who have initiated olaparib within the last two months of study entry, or for whom the decision to be treated with olaparib has been made by their physician
* Who have been informed and are not opposed to this data collection

Exclusion Criteria:

* Patients opposed to the collection of their data
* Patients participating in a clinical trial with an investigational prostate cancer targeted drug within 30 days prior to Olaparib initiation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male patients with metastatic castration-resistant prostate cancer who have initiated olaparib or for whom the decision to be treated with olaparib has been made by their physician.
  A sample of approximately 300 patients is expected to be enrolled from around 60 french sites.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2028-10-13 (Estimated); Study Completion 2028-10-13 (Estimated)

PRIMARY OUTCOMES:
Time to treatment discontinuation (TTD) | Up to 36 months from olaparib initiation
  TTD is defined as the time from the first day of olaparib treatment to the day that olaparib stopped for whatever reason or the date of death due to any cause, whichever comes first

CONTACTS AND LOCATIONS:
Locations (47):
- France (47):
  - Research Site, Amiens
  - Research Site, Angers
  - Research Site, Antony
  - Research Site, Argenteuil
  - Research Site, Avignon
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Challes-les-Eaux
  - Research Site, Chambray-lès-Tours
  - Research Site, Champigny-sur-Marne
  - Research Site, Clermont-Ferrand
  - Research Site, Compiègne
  - Research Site, Créteil
  - Research Site, Epagny METZ Tessy
  - Research Site, Ermont
  - Research Site, FORT de France
  - Research Site, Fréjus
  - Research Site, Grenoble
  - Research Site, Le Chesnay
  - Research Site, Le Coudray
  - Research Site, Le Mans
  - Research Site, Levallois-Perret
  - Research Site, Lyon
  - Research Site, Mantes-la-Jolie
  - Research Site, Marseille
  - Research Site, Morlaix
  - Research Site, Nancy
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, ORL ANS
  - Research Site, Paris
  - Research Site, Pointe à Pitre
  - Research Site, Poitiers
  - Research Site, Pontoise
  - Research Site, Quint-Fonsegrives
  - Research Site, Rouen
  - Research Site, Saint Denis- LA Reunion
  - Research Site, Saint-Doulchard
  - Research Site, Saint-Etienne
  - Research Site, Saint-Grégoire
  - Research Site, Saint-Mandé
  - Research Site, Saint-Nazaire
  - Research Site, Strasbourg
  - Research Site, Suresnes
  - Research Site, Tours
  - Research Site, Vannes
  - Research Site, Vantoux